CLINICAL TRIAL: NCT07353580
Title: Impact of Selective Curettage and Tissue Adhesive on the Clinical Outcomes of Endodontic Microsurgery: A Randomized Controlled Trial
Brief Title: Selective Curettage and Tissue Adhesive in Endodontic Microsurgery
Acronym: Microsurgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Adel El-Dreny Mohamed, Assistant Lecturer, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A02010024 RC
Record Dates: First submitted 2026-01-07; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Healing and Patient Related Outcomes
MeSH Terms: interventions — Sutures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Complete Periapical Lesion Curettage and Suturing (Active Comparator): patients underwent conventional endodontic microsurgery with complete removal of the periapical lesion followed by flap repositioning and closure using sutures.
  Interventions: Procedure: Complete Periapical Lesion Curettage and Suturing
- Selective Lesion Curettage and Cyanoacrylate Tissue Adhesive (Experimental): Patients underwent endodontic microsurgery with selective removal of approximately 40-70% of the periapical lesion, followed by flap closure using cyanoacrylate tissue adhesive without sutures.
  Interventions: Procedure: Selective Lesion Curettage and Cyanoacrylate Tissue Adhesive

INTERVENTIONS:
Procedure: Selective Lesion Curettage and Cyanoacrylate Tissue Adhesive — Selective curettage is a conservative approach to treat periapical lesions by removing part of the granulomatous tissue while avoiding complications and damage to the neighboring structures. It also provides the least traumatic approach with minimal post-operative complications. It had an additional advantage, which is providing tissue samples for biopsy of the lesion, especially in cases where there was a diagnostic dilemma regarding its origin . In the selective curettage technique, approximately 50-70% of the granulomatous tissue was removed while preserving the portion in close proximity to critical areas, followed by standard root-end resection and retrofilling then Clinical and radiographic assessments, including CBCT, for bone healing assesment .
  Arms: Selective Lesion Curettage and Cyanoacrylate Tissue Adhesive
Procedure: Complete Periapical Lesion Curettage and Suturing — Complete Periapical Lesion Curettage and Suturing is a conventional endodontic microsurgical procedure performed to manage persistent periapical pathology following root canal treatment. After administration of local anesthesia, a full-thickness mucoperiosteal flap is elevated to expose the periapical region. The periapical lesion is completely curetted and removed, followed by apical root-end resection. A retrograde cavity is prepared using ultrasonic tips and sealed with a biocompatible root-end filling material. Hemostasis is achieved, and the surgical flap is repositioned and stabilized using conventional sutures. This approach represents the standard surgical protocol for endodontic microsurgery and serves as the active comparator in this study.
  Arms: Complete Periapical Lesion Curettage and Suturing

SUMMARY:
The goal of this randomized clinical trial is to determine whether selective curettage combined with cyanoacrylate tissue adhesive improves clinical outcomes in endodontic microsurgery compared with the conventional approach. The study purpose is to evaluate the postoperative healing associated with this conservative surgical protocol.

The main questions it aims to answer are:

Does selective curettage with tissue adhesive reduce postoperative pain, swelling, and complications compared to complete curettage with suturing?

How does selective curettage affect clinical and radiographic healing of persistent periapical lesions?

Researchers compared complete lesion curettage with suturing to selective curettage (40-70% lesion removal) with cyanoacrylate tissue adhesive closure to assess differences in healing and patient-related outcomes.

Participants :

Underwent endodontic microsurgery using one of the two surgical protocols Attended follow-up visits at 1, 3, and 7 days for clinical evaluation of pain, swelling ,Discomfort , Bleeding , Local reaction and Wound Dehiscence

Attended follow-up visits at 3, 6, and 12 months for clinical and radiographic evaluation of periapical healing using 2D radiographs and CBCT

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and older consenting to the surgical procedure as well as agreeing to preoperative and at least 1 follow-up CBCT evaluation.
2. Noncontributory medical history (American Society of Anesthesiologists class I, II).
3. Teeth with periapical lesions that had been previously treated or retreated but symptoms persist or recurrent.
4. Radiographic presence of true endodontic lesion close to vital critical structure.

Exclusion Criteria:

1. Nonconsenting patients and patients younger than 18 years of age.
2. Medical history with the American Society of Anesthesiologists class III to V.
3. Insufficient coronal restoration.
4. Nonrestorability or traumatized teeth.
5. Mobility > 1.
6. Vertical root fracture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-12-25 (Actual); Primary Completion 2026-01-29 (Estimated); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | (1st, 3rd, and 7th day post-operative)
  Pain intensity is assessed using the Visual Analogue Scale (VAS, 0-10)
Swelling | 1st, 3rd, and 7th day post-operative
  Presence of swelling is assessed clinically by visual inspection and physical examination and recorded as a binary outcome (present / absent)

SECONDARY OUTCOMES:
Bleeding | 1st, 3rd, and 7th day post-operative
  Post-operative bleeding presence is assessed as a binary outcome (Yes / No)
Radiographic Bone healing | 3, 6 , and 12 months
  Radiographic bone healing is assessed using standardized periapical radiographs (2D) and cone beam computed tomography (CBCT, 3D)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A El-dreny, Assis.Lec, Principal Investigator — Faculty of Dentistry , Mansoura University
Locations (1):
- Faculty of Dentisrty , Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nesari R, Kratchman S, Saad M, Kohli MR. Selective Curettage: A Conservative Microsurgical Approach to Treating Large and Complicated Lesions. J Endod. 2020 Nov;46(11):1782-1790. doi: 10.1016/j.joen.2020.07.023. Epub 2020 Jul 29. PMID 32738339